CLINICAL TRIAL: NCT04181905
Title: The Relationship Between Kinesiophobia, Physical Activity Level and Quality of Life in Asthma Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Other Study IDs: 21.02.2019/35
Record Dates: First submitted 2019-11-27; First posted 2019-12-02 (Actual); Last update posted 2020-09-11 (Actual); Status verified 2019-11

CONDITIONS: Asthma
Keywords: Asthma, Kinesiophobia, Physical Activity, Quality of Life
MeSH Terms: conditions — Asthma; Kinesiophobia; Motor Activity | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire — Firstly, demographic information (name-surname, date of birth, gender, age, height, body weight, dominant hand, family structure, social security, educational status, occupation, smoking, alcohol use, assistive device drug use, resume, surname, complaints). Data collection tools will then be applied to patients by face to face interview technique. Evaluation of kinesiophobia Assessment of quality of life in asthma patients with TAMPA questionnaire Assessment of physical activity level with Asthma Quality of Life Questionnaire (AQLQ) Assessment of physical activity level with International Physical Activity Questionnaire-Short Form (IPAQ) is planned.

SUMMARY:
Asthma is a heterogeneous disease characterized by chronic airway inflammation characterized by time-varying respiratory symptoms such as wheezing, shortness of breath, chest tightness and cough, with limitation of expiratory airflow. These variations are often triggered by exercise, exposure to allergens or an irritation, weather changes or viral respiratory diseases (Karakış, 2018). Increased respiratory distress decreases the patient's activity, decreases the condition and makes the individual dependent in daily life. In the studies conducted in asthma patients, the cases stated that they perceived their illness as an obstacle against physical activity and thus they were pushed to immobility (Kırtay & Oğuz, 2011). In the literature, no study on the variable of kinesiophobia in asthma was found. The aim of this study was to investigate the relationship between kinesiophobia and physical activity level and quality of life in asthma patients.

DETAILED DESCRIPTION:
Asthma is a chronic inflammatory disease characterized by increased airway sensitivity to various stimuli and reversible airway obstruction (Soyuer et al., 2013). Bronchial hypersensitivity associated with chronic airway inflammation causes wheezing, dyspnea, chest tightness, and cough attacks, especially at midnight or morning. These attacks are associated with varying degrees of airway obstruction and usually improve with treatment or spontaneously (Arslan, 2011). Three mechanisms are responsible for the pathogenesis of asthma. These include reversible airway obstruction, airway inflammation, and increased airway sensitivity (Soyuer et al., 2013). Although it is known that genetic and environmental factors play a role in asthma formation, etiopathogenesis has not been fully explained (Arslan, 2011). Approximately 300 million people worldwide suffer from asthma and this prevalence increases by 50% every ten years. Hospitalization is frequently seen in patients with asthma (Autumn, 2015). It is estimated that approximately 250,000 people die annually due to asthma. No relationship was found between prevalence and mortality (Autumn, 2015). Asthmatic patients have intermittent symptoms such as wheezing, dyspnea, chest tightness, and dry cough. Stimulants such as allergens, air pollution, gastroesophageal reflux, stress and exercise cause these symptoms. 90% of untreated asthmatics develop asthma symptoms during exercise (Dursun et al., 2013). Airway obstruction due to exercise occurs in 40-90% of asthmatics, decreases the ability to exercise and patients prefer a more sedentary lifestyle. Patients with asthma have low physical activity levels because they avoid exercising due to anxiety and depression, inactivity, fatigue, dyspnea (Autumn, 2015). The ability to perform activities and the ability to perform daily living activities are components of quality of life. In many studies, it has been found that quality of life is affected in individuals with chronic lung disease. Quality of life can be assessed with many disease-specific questionnaires. Asthma patients experience problems in many areas in terms of quality of life, including day and night disease symptoms, impaired daily living activities, and reduced quality of life. Asthma is associated with decreased quality of life and morbidity. Asthma symptoms reduce performance at school and at work; affects learning and reduces quality of life. It is stated that asthma has a negative effect on quality of life, physical, physiological and social function (Autumn, 2015).

Airway obstruction due to exercise decreases physical activity in asthmatic patients. This may give rise to fear of movement over time. Avoidance of movement is called kinesiophobia. Kinesiophobia is a condition that occurs when patients want to perform their previous functions, especially in chronic painful disease processes.

Kinesiophobia is an avoidance phenomenon within the cognitive behavioral avoidance model and patients may limit their activity in daily life in case of symptoms of deterioration or the occurrence of symptoms. This may result in emotional problems and life dissatisfaction in later periods (Yumin et al., 2017). Kinesiophobia has been the subject of study in cardiopulmonary cases, but there is no research on kinesiophobia in asthma. In this study, the effect of kinesiophobia on physical activity level and quality of life in asthma will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Being 18-65 years old T
* Turkish reading, writing, understanding
* Volunteering to participate in the research

Exclusion Criteria:

* Having communication problems, not being cooperative, having a psychiatric diagnosis or using medication
* Severe comorbid diseases (heart, respiratory, gastrointestinal, neurological diseases) that may cause movement limitation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population of the study was the patients diagnosed with asthma. The sample is planned to be composed of 40 people who meet the criteria of reading, read the information form and signed the informed consent form.
Sampling Method: Probability Sample
Enrollment: 42 (Estimated)
Dates: Start 2019-04-21 (Actual); Primary Completion 2020-12-18 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
Tampa Kinesiophobia Scale (TSK) | 7 days
  The Tampa Scale of Kinesiophobia (TSK) that was developed in 1990 is a 17 item scale originally developed to measure the fear of movement related to chronic lower back pain. The TSK consists of 17 questions.A score of 17 is the lowest possible score, and indicates no kinesiophobia or negligible. A score of 68 is the highest possible score and indicates extreme fear of pain with movement.
International Physical Activity Questionnaire Short Form (IPAQ-SF) | 7 days
  The International Physical Activity Questionnaire short-form (IPAQ-SF) is one of the most widely used self-report questionnaires to assess PA. IPAQ-SF is a self-report questionnaire that assesses PA in the last 7 days [9-10]. Using the IPAQ-SF scoring system, the total number of days and minutes of PA were calculated for each participant as recommended in the IPAQ website [32]. The IPAQ-SF records the activity in four intensity levels: sitting, walking, moderate intensity (e.g., leisure cycling), and vigorous intensity (e.g, running or aerobics). MET method was used to determine the level of physical activity. Standard values for these activities were established. The generated values are expressed as follows; Severe Physical Activity = 8.0 MET, Moderate Severe Physical Activity = 4.0 MET, Walking = 3.3 MET, Sitting = 1.5 MET. Using these values, daily and weekly physical activity levels are calculated.
Asthma Quality of Life Questionnaire (AQLQ) | 14 days
  The Asthma Quality of Life Questionnaire (AQLQ) was developed to measure the functional problems (physical, emotional, social and occupational) that are most troublesome to adults (17-70 years) with asthma. Participants were asked to score the importance of each of the positively identified problems (0= not important - 4 = very important). The highest scoring problems were the same for both men and women, for patients with a wide range of asthma severity (no medication to oral steroids) and in different age groups.

CONTACTS AND LOCATIONS:
Overall Officials: Aysel Yildiz Ozer, Study Chair — Marmara University, Department of Physiotherapy and Rehabilitation; Seda Karaca, Principal Investigator — Marmara University, Department of Physiotherapy and Rehabilitation
Locations (2):
- Turkey (Türkiye) (2):
  - Marmara University, Istanbul
  - Seda Karaca, Istanbul

IPD SHARING:
Plan to Share IPD: No